

7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

Ab interno Gelatin Stent with mitomycin C using targeted supra-tenon's placement

PI: Iqbal Ike K Ahmed MD FRCSC

Research Staff: Fady Sedarous

Study Coordinator: Ayda Shahidi

Version 1.0

Dec 14th, 2018



7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

### Table of Abbreviations

Any abbreviations that you will be using in your protocol <u>must</u> be defined in this table in alphabetical order. If no abbreviations are being used, then this section does not need to be included

GVT—Gelatin Stent vs. Trabeculectomy

MMC—Mitomycin C

IOP—Intraocular Pressure

PKP—Penetrating Keratoplasty

DALK—Deep Anterior Lamellar Keratoplasty

DSAEK—Descemet's stripping automated endothelial keratoplasty

DMEK—Descemet's membrane endothelial keratoplasty

CPC—Cyclophotocoagulation

AC—Anterior Chamber

POM—Post-op month



7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

### Background

The Xen-45 gelatin microstent (Allergan, Dublin, Ireland) is a novel, bleb-forming microinvasive glaucoma surgery (MIGS).¹ Creation of a filtering bleb through the gel stent and under the conjunctiva lowers intraocular pressure (IOP) by bypassing the natural outflow pathway of aqueous. A recent retrospective cohort study showed comparable safety and risk of failure to trabeculectomy.² Amongst the main advantages of this device is the ability to create a bleb without dissecting and disrupting tissue, thus decreasing the amount of wound healing and potentially limiting bleb failure. However, despite demonstrating similar efficacy and safety to trabeculectomy,² the Xen-45 gelatin microstent continues to suffer from occasional surgical failure due to fibrosis of the filtering bleb, and obstruction of the stent.³ Although antimetabolites, such as mitomycin C, have decreased reactionary wound healing that can result following surgery, fibrosis may still occur, especially when the components of the Xen-45 gelatin microstent are in close proximity to the fibroblastic structures of tenon's fascia.⁴,5

Tenon's capsule resembles a sponge-like layer with multiple adhesions to the overlying conjunctiva and underlying episclera. Implantation of the XEN within this space creates a higher risk of obstruction and subsequent failure. To ensure the lowest potential for occlusion, bleb scarring, and failure, one must ensure careful placement of the device in the subconjunctival space, avoiding intra-tenon's placement. Placement in the supra-tenon's space is believed to maximize aqueous outflow, while preventing obstruction, limiting fibrosis of the bleb, and promoting long-term patency. Despite the theoretical merits, long-term data of outcomes after targeted supra-tenon's placement is needed to fully assess its potential in improving Xen-45 microstent outcomes.

### Research Question/Objective

#### Hypothesis

• Targeted supra-tenon's placement of the Xen-45 gel microstent results in higher success, less needling and lower IOPs than non-targeted placement.

#### Primary objective

• Evaluate outcomes of patients receiving an ab interno gelatin stent with mitomycin C (MMC) using targeted supra-tenon's placement to patients receiving an ab interno gelatin stent with non-targeted placement.

# prism Pre INSTITUTE

#### **BRAMPTON**

7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

#### Secondary objectives

- Intraoperative complications: corneal abrasion or perforation, hyphema, subconjunctival bleeding, gelatin stent fracture or need for re-implanation, iris prolapse, suprachoroidal hemorrhage, vitreous loss or posterior capsule rupture.
- Management interventions (not considered complications): bleb needling, AC reformation, suture release, digital ocular compression, use of glaucoma medications, or laser/tpa to blocked ostomy or lumen.
- IOP: mean IOP, mean decrease in IOP from baseline, IOP thresholds of ≥6 and ≤17, ≥6 and ≤14, and ≥6 and ≤21 (mmHg).
- Vision: number of patients who lose more than two lines of best corrected visual acuity, post-operative cataract surgery rates, auto-refraction.
- Glaucoma medications: number of topical glaucoma medications and percentage of patients on glaucoma medications.
- Visual recovery: percentage of patients who achieve baseline best corrected visual acuity at 1 week, 1 month, 3 months, and annually thereafter.
- Non-protocol visits: number of non-scheduled non-protocol visits.

#### Aim of the project

• Retrospectively obtain data through a chart review for exploratory purposes.

### Study Design

#### Population + Recruitment Strategies

- Patients aged 30-90 with primary or pigmentary/pseudoexfolliative open angle, primary closed angle, or combined mechanism glaucoma with IOP of 18-40 mmHg on maximum tolerated medical therapy who received a gelatin stent with MMC at Prism Eye Institute from June 2012 to August 2019.
- Exclusions: other forms of glaucoma, prior incisional glaucoma surgery, CPC, prior corneal graft (PKP, DALK, DSAEK, DMEK).

Sample Size



7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

• Assuming an alpha of 0.05, a clinically significant IOP difference of 3 mmHg and a standard deviation of 5 mmHg, the estimated sample size is 88 eyes (44 eyes per group).

#### Tools for Data Collection

• Data will be collected from the Electronic Medical Record.

Methodology

#### **Outcome:**

Survival analysis will be determined by the following success/failure criteria:

#### 1. Complete success:

- a. IOP: 6-17 mmHg and on no glaucoma medications (starting after POM1[3]) at least 1 month after surgery with no reoperation.
- b. Absence of the following complications:
  - Starting after POM1[3]: shallow AC w/ iridocorneal touch, any hyphema, corneal edema, wound leak/dehiscience, choroidal effusion, malignant glaucoma, dellen/non-healing epithelial defect, ptosis, diplopia.
  - ii. At any point: additional glaucoma surgery, loss of light perception vision, vitreous hemorrhage, ≥2mm hyphema, hypotony maculopathy, implant migration/blockage/exposure/extrusion, macular edema, choroidal effusion/hemorrhage requiring drainage, suprachoroidal hemorrhage, retinal detachment, suture abscess/blebitis/endophthalmitis
- c. Stable functional testing
  - After POM1[3] no decrease in best corrected visual acuity of more than 2 lines from baseline on 2 consecutive visits (unless deemed to be due to corneal or retinal disease—e.g., retinal vein occlusion)

#### 2. Qualified success:

a. 'Complete success' criteria except that IOP can be above IOP thresholds, and then reduced to within the 'Complete criteria' by medications or laser in 3 visits or less.

<u>Statistical Analysis:</u> Analysis of variance (ANOVA) and Wilcoxon signed-rank test will be used to compare univariate normal and non-normal continuous baseline characteristics and outcomes. Fisher exact tests will be used to compare univariate categorical baseline characteristics and outcomes. Time to failure will be defined as the time from surgery to the patient no longer meeting the 'success' criteria. Multivariate analysis will be performed with Cox proportional hazard regression analysis. A p-value of 0.05 or less will be considered statistically significant.

## prism eye institute

#### **BRAMPTON**

7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

#### Safety Considerations

• Given the nature of this project (retrospective chart review) there are no safety considerations.

#### Data Analysis

• Data analysis will follow the plan outlined above and use SAS Studio (Cary, NC).

#### Perceptions of Bias

- Information bias: Neither the patients nor clinicians are masked, thus in theory reporting can be influenced by performance bias and clinician beliefs. This is an inherent limitation of a retrospective study. The use of objective clinical measures to quantify success minimizes this bias.
- There may be differential loss to follow-up in the study. Patients can be lost to follow-up for a variety of reasons: because they are doing well (sent back to the referring physician), not doing well (had a complication and have sought a second opinion), or lost to follow-up for other reasons not influenced by outcomes.

#### Follow-up

• The follow-up will be according to the patient's electronic health record.

### **Project Feasibility**

#### Ethical considerations

• Given the retrospective nature of this project the main concern is the protection of the personal health information of the patients studied. The data will be collected without personal identifying information (instead using a unique identifier), and published will be in aggregate as to not reveal personal information about any patient in an identifiable manner.

# prism eye institute

#### **BRAMPTON**

7700 Hurontario St, Unit 605, L6Y 4M3

#### **MISSISSAUGA**

3200 Erin Mills Pkwy, Unit 1, L5L 1W8 71 King Street West, Unit 207, L5B 4A2

### References

- 1. Conlon R, Saheb H, Ahmed IIK. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017;52(1):114-124. doi:10.1016/j.jcjo.2016.07.013.
- 2. Schlenker MB, Gulamhusein H, Conrad-Hengerer I, et al. Efficacy, Safety, and Risk Factors for Failure of Standalone Ab Interno Gelatin Microstent Implantation versus Standalone Trabeculectomy. In: Ophthalmology.; 2017. doi:10.1016/j.ophtha.2017.05.004.
- 3. Fea AM, Spinetta R, Cannizzo PML, et al. Evaluation of Bleb Morphology and Reduction in IOP and Glaucoma Medication following Implantation of a Novel Gel Stent. J Ophthalmol. 2017. doi:10.1155/2017/9364910.
- 4. Ca C, Wang J, Hau S, Htoon HM, Barton K. Original Article XEN-45 collagen implant for the treatment of uveitic glaucoma. Clin Exp Ophthalmol. 2018;46(October 2017):339-345. doi:10.1111/ceo.13087.
- Crowston JG, Akbar AN, Constable PH, Occleston NL, Daniels JT, Khaw PT.
  Antimetabolite-induced apoptosis in Tenon's capsule fibroblasts. Investig Ophthalmol Vis Sci. 1998.
- 6. Kakizaki H, Takahashi Y, Nakano T, et al. Anatomy of Tenons capsule. Clin Exp Ophthalmol. 2012. doi:10.1111/j.1442-9071.2011.02745.x.
- 7. Lewis RA. Ab interno approach to the subconjunctival space using a collagen glaucoma stent. J Cataract Refract Surg. 2014;40(8):1301-1306. doi:10.1016/j.jcrs.2014.01.032.